CLINICAL TRIAL: NCT06982651
Title: A Randomized, Double-Blind, Placebo-Parallel-Controlled Phase Ⅰ Clinical Trial of the Tolerability, Safety, Pharmacokinetics and Food Effects of MI078 Capsules in Single and Multiple Doses in Healthy Chinese Subjects
Brief Title: A Study on the Safety, Pharmacokinetics, and Food Effects of MI078 Capsules
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nanjing Minova Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 23090
Record Dates: First submitted 2025-04-24; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-03

CONDITIONS: Postpartum Depression
Keywords: Postpartum Depression; MI078; Minova
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MI078 capsule (Experimental): MI078 capsule
  Interventions: Drug: MI078
- placebo (Placebo Comparator): Placebo of MI078 Capsule
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MI078 — Dosage Form: Capsule Specification: 25 mg Administration and Dosage: Oral. 1 capsule per dose, once daily. Duration of Treatment: 1 day
  Dosage Form: Capsule Specification: 50 mg Administration and Dosage: Oral. 1 capsule per dose, once daily. Duration of Treatment: 1 day
  Dosage Form: Capsule Specification: 200 mg
  Administration and Dosage: Oral. Options include:
  * 1 capsule per dose, once daily;
  * 2 capsules per dose, once daily;
  * 3 capsules per dose, once daily;
  * 4 capsules per dose, once daily; Duration of Treatment: 1 day .
  Dosage Form: Capsule Specification: 200 mg
  Administration and Dosage: Oral. Options include:
  * 1 capsule per dose, twice daily;
  * 2 capsules per dose, twice daily; Duration of Treatment: 7 days .
  Dosage Form: Capsule Specification: 50mg
  Administration and Dosage: Oral. Options include:
  - 5 capsule per dose, Three times a day Duration of Treatment: 3 days .
  Arms: MI078 capsule
Drug: Placebo — Placebo of MI078 Capsule
  Arms: placebo

SUMMARY:
This study was divided into three studies, namely, a single administration study, a food impact study, and a multiple administration study.

DETAILED DESCRIPTION:
Single-dose study：Eight single-dose cohorts (25 mg, 50 mg, 100 mg, 200 mg, 400 mg, 600 mg, 800 mg, and 1000mg) were planned, as described in the table below. In the first and second dose groups (25 mg and 50 mg), a single oral dose of MI078 capsules was given to 1 male and 2 females in a single-center, open-label design. The tolerance and safety of MI078 capsules were evaluated. Dose groups 3-8 were designed in a single-center, randomized, double-blind, placebo-controlled design. Each dose group was planned to enroll 8-10 volunteers, half male and half female (see the table below for details). On the basis of PK and safety data, the actual dose escalation could be adjusted accordingly.

Food Impact Studies：This study adopted a randomized, open, two-sequence, two-cycle crossover design, and the 400 mg dose was selected for the food impact test. Fourteen healthy volunteers, both male and female, were randomly divided into two sequence groups according to the fasting - postprandial and postprandial - fasting administration methods. Each sequence group had 7 volunteers and was divided into two cycles. All volunteers were required to be hospitalized from 1 day before administration to 72 h after administration (day 4). During this hospitalization, volunteers were required to complete the collection of pharmacokinetic samples (blood samples, collection to 72 h after administration). All volunteers could be discharged after the collection of the above biological samples and the corresponding safety assessment. After a washing period of at least 7 days, the second cycle of PK test could be carried out. The collection of PK blood samples and the corresponding safety check in the second cycle were the same as those in the first cycle.

Multiple dosing studies：The multiple-dose study was a single-center, multi-dose, randomized, double-blind, placebo-controlled design. A total of 30 healthy volunteers (half male and half female) were planned to be enrolled. When the higher-dose arm of the single-dose study had been evaluated for tolerability, the multiple-dose study with a sublower dose could proceed. The dose for this study could be adjusted to 250mg for group 3 based on safety and PK data (blinded) from the completed study results (200mg and 400mg groups). MI078 capsules or placebo were administered to 10 volunteers in each of three dose cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Are willing and able to provide signed informed consent to participate in the study and to comply with all study procedures and scheduled visits.
* Are an adult aged 18 to 45 years, inclusive.
* Have a BMI between 19.0 and 26.0 kg/m² (inclusive of boundary values) and weigh ≥50.0 kg if male, or ≥45.0 kg if female.
* Have a total score for suicidal ideation ≤12 points and a score for the dissimulation factor <4 points on the suicide risk assessment scale at the time of screening.
* Have regular menstrual cycles, occurring within 28 ± 7 days (female volunteers only).
* Have had a depressive episode that began no earlier than the third trimester and no later than the first 4 weeks following delivery (if applicable).
* Are ≤9 months postpartum at Screening (if applicable).

Exclusion Criteria:

* Have a history or current diagnosis of any clinically significant diseases of the cardiovascular, endocrine, nervous, digestive, respiratory, urinary, and reproductive systems, hematology, immunology, psychiatry, or metabolic abnormalities, or any other diseases that may interfere with the study results.
* Have a family history of risk factors for torsades de pointes, or a history of short QT syndrome, long QT syndrome, unexplained sudden death or drowning in young age (≤40 years), or sudden infant death syndrome in first-degree relatives (i.e., biological parents, siblings, or children).
* Are engaged in high-altitude work or other occupations involving hazardous mechanical operations.
* Have a history of allergies to drugs, food, or other substances.
* Have experienced vomiting within 24 hours before dosing, which is assessed by the investigator to affect the study or impact the safety of the volunteer.
* Have undergone surgery within 4 weeks before the study or are planned to undergo surgery during the study period.
* Have taken any medications or health supplements (including traditional Chinese medicine) within 14 days before the study.
* Have used any drugs that inhibit or induce hepatic drug metabolism within 30 days before the study (e.g., inducers-barbiturates, carbamazepine, phenytoin, corticosteroids, omeprazole; inhibitors-SSRI antidepressants, cimetidine, diltiazem, macrolides, nitroimidazoles, sedative-hypnotics, verapamil, fluoroquinolones, antihistamines).
* Have participated in any clinical trial and taken any investigational drug within 3 months before the study.
* Have donated blood or experienced significant blood loss (≥200 mL, excluding menstrual blood loss in women), received blood transfusions, or used blood products within 3 months before enrollment.
* Are pregnant or breastfeeding, or cannot use one or more non-pharmacological contraceptive methods during the study period.
* Have special dietary requirements that prevent them from adhering to the standardized diet.
* Consume excessive amounts of tea, coffee, and/or caffeine-containing beverages (more than 8 cups per day, 1 cup = 250 mL).
* Have consumed excessive amounts of citrus-rich beverages or foods (e.g., grapefruit, oranges) within 48 hours before the first admission to the ward.
* Are smokers or have smoked more than 5 cigarettes per day within 3 months before the study or cannot refrain from using any tobacco products during the study.
* Are alcohol abusers or have regularly consumed alcohol within 6 months before the study (i.e., more than 14 units of alcohol per week, 1 unit = 360 mL of beer or 45 mL of 40% spirits or 150 mL of wine) or cannot refrain from using any alcohol-containing products during the study.
* Are drug abusers or have used soft drugs (e.g., marijuana) within 3 months before the study or hard drugs (e.g., cocaine, phencyclidine) within 1 year before the study.
* Have abnormal vital signs (systolic blood pressure <90 mmHg or >140 mmHg, diastolic blood pressure <50 mmHg or >90 mmHg; pulse rate <50 bpm or >100 bpm, respiratory rate <12 breaths per minute or >20 breaths per minute) or abnormal physical examination, electrocardiogram (normal ECG requirements: male QTcF ≤450 ms, female QTcF ≤470 ms; PR interval ≤200 ms; QRS complex duration ≤120 ms), or laboratory tests with clinically significant abnormalities (as judged by the clinical research physician).
* Have positive results for hepatitis B surface antigen, hepatitis C antibody, preliminary screening for HIV antigen/antibody, or syphilis serological reaction.
* Have difficult venous blood collection or a history of needle fainting or blood fainting, who are deemed unsuitable for enrollment by the investigator.
* Are likely to be unable to complete the study for other reasons or are deemed ineligible by the investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 98 (Actual)
Dates: Start 2023-09-09 (Actual); Primary Completion 2024-03-18 (Actual); Study Completion 2024-03-18 (Actual)

PRIMARY OUTCOMES:
Incidence, severity, and causality of AEs, SAEs | up to 72 hours after the last dose
  Clinical safety assessments will be conducted for all spontaneously reported and directly observed adverse events (AEs) and serious adverse events (SAEs). AEs should also include abuse-related AEs (such as insomnia, sedation, hallucinations, tremors, and dissociative states) and withdrawal reactions (including headache, anxiety, nausea, vomiting, tremors, decreased attention, irritability, anger, and sleep disturbances).
vital signs | up to 72 hours after the last dose
  Any abnormal changes in vital signs
SpO₂ | up to 72 hours after the last dose
  Any abnormal changes in SpO₂ (peripheral capillary oxygen saturation)
12-lead electrocardiogram (ECG) | up to 72 hours after the last dose
  HR, RR interval, PR interval, QRS complex duration，QTcF=QT/(RR^0.33)
Modified Observer's Assessment of Alertness and Sedation Scale（MOAA/S） | up to 72 hours after the last dose
  MOAA/S scale is a validated 6-point scale assessing the responsiveness of patients, coinciding with the American Society of Anesthesiologists (ASA) continuum of sedation。The scale rates patient responsiveness as follows： 5：Responds readily to name spoken in normal tone 4：Lethargic response to name spoken in normal tone 3：Responds only after name is called loudly and/or repeatedly 2：Responds only after mild prodding or shaking
  1：Responds only after painful trapezius squeeze 0：Does not respond to painful trapezius squeeze
Stanford Sleepiness Scale (SSS) | up to 72 hours after the last dose
  The Stanford Sleepiness Scale (SSS) is a widely used self-assessment tool designed to measure subjective levels of sleepiness or alertness. It consists of a 7-point scale that allows individuals to rate their current level of alertness or sleepiness. The scale is as follows:
  1. Feeling active, vital, alert, or wide awake
  2. Functioning at a high level, but not at peak; able to concentrate
  3. Awake, but relaxed; responsive but not fully alert
  4. A little foggy; not at best
  5. Foggy; losing interest in remaining awake; slowed down
  6. Sleepy, woozy, fighting sleep; prefer to lie down
  7. No longer fighting sleep, sleep onset soon; having dream-like thoughts

SECONDARY OUTCOMES:
Plasma Concentrations of MI078 | up to 72 hours after the last dose
  PK Parameters of MI078 will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Third Xiangya Hospital, Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No